CLINICAL TRIAL: NCT04709458
Title: A Phase I Study to Assess the Safety and Early Efficacy of TBX-2400 in Enhancing Engraftment in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant for the Treatment of Acute Myelogenous Leukemia or Myelofibrosis
Brief Title: Safety and Early Efficacy Study of TBX-2400 in Patients With AML or Myelofibrosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taiga Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBX-2400-001
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Myelofibrosis; Acute Myelogenous Leukemia
Keywords: Myelofibrosis; Leukemia; Allogeneic stem cell transplant; Acute Myelogenous Leukemia; Myeloproliferative disorders; Primary myelofibrosis; Bone Marrow Cancer; Bone Marrow Transplant; Acute Myeloid Leukemia
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myeloid, Acute; Leukemia; Myeloproliferative Disorders; Bone Marrow Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TBX-2400 treatment (Experimental): Single intravenous infusion of TBX-2400
  Interventions: Biological: TBX-2400

INTERVENTIONS:
Biological: TBX-2400 — Hematopoietic stem cells transplantation

SUMMARY:
This is a study of allogeneic stem cell transplantation with TBX-2400 in adult subjects with Acute Myelogenous Leukemia (AML) or Myelofibrosis (MF).

The donor cells are exposed to a protein that has been shown in the laboratory to improve the ability of the donor cells to make blood and immune cells after transplant. Exposure of the donor cells to this protein does not modify the genes in the cells in any way.

This study has two goals. The first goal is to find out if transplant with TBX-2400 is safe. The second goal is to find out what effects TBX-2400 stem cells have on time to engraftment in adult subjects with AML or MF.

The study hypothesis is that TBX-2400 cells will shorten the time to immune reconstitution after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. For crAML: AML with ≥5% blasts (either by morphology or by multi-parameter flow cytometry [MFC]) in a marrow aspirate obtained within 21 days of enrollment in the trial, and following the administration of at least two prior courses of chemotherapy;
2. For MF: primary MF or MF that has progressed from a myeloproliferative disease. Dynamic International Prognostic Scoring System (DIPSS)-plus to be utilized to support the inclusion of MF subjects at screening;
3. Subject undergoing allogeneic stem cell transplantation on the decision of transplanting physician;
4. Signed informed consent of donor and recipient;
5. Subjects of ≥ 18 years of age (no upper age limit);
6. Donor agrees to donate bone marrow-derived or mobilized peripheral blood stem cells;
7. Subjects with Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2;
8. Adequate pulmonary function with Diffusing Capacity for Carbon Monoxide (DLCO) > 50;
9. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception (e.g. sterilization, hormone implants, hormone injections, intrauterine devices, or vasectomized partner with combined use of condom and/or birth control pills) from screening until 6 months after TBX-2400 transplantation;
10. Able to adhere to all trial treatments and procedures.

Exclusion Criteria:

1. Previous stem cell transplantation;
2. For MF: Blasts > 10% in a marrow aspirate obtained within 30 days of screening;
3. Renal function: serum creatinine > 1.5 x Upper Limit of Normal (ULN);
4. Hepatic function: impaired synthetic function as indicated by a serum fibrinogen below the normal limit. Aspartate transaminase/alanine transaminase (AST/ALT) > 3.0 x ULN. Bilirubin, > 1.5 x ULN;
5. Cardiac function: ejection fraction < 45% as determined by echocardiography;
6. Prior malignancy active within previous three years - except for locally curable cancers such as cutaneous basal or squamous cell cancer, superficial bladder cancer, carcinoma in situ of cervix or breast, or carcinoma in situ of the prostate;
7. Positive pregnancy test or breastfeeding for women of childbearing age;
8. Serologic evidence of chronic Hepatitis B virus infection or Hepatitis C exposure;
9. Known history of positive test for Human Immunodeficiency Virus (HIV) or known Acquired Immunodeficiency Syndrome (AIDS);
10. Hypersensitivity to any trial medication (including the preparative regimen, TBX-2400 treatment and any prophylaxis or other medication planned);
11. Presence of a serious or uncontrolled medical disorder that, in the opinion of the Investigator, may increase the risk associated with trial participation or trial drug administration, impair the ability of the participant to receive protocol therapy, or interfere with interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-08-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events according to NCI-CTCAE Version 5.0 | Two years
  Adverse events from subject reporting or other assessments
Transplant engraftment | 1 year
  Assessment of transplant engraftment will include absolute neutrophil count, untransfused platelet count and donor chimerism

SECONDARY OUTCOMES:
Immune reconstitution as measured by CD3+ cell count | Up to Day 360
  Immune reconstitution as measured by CD3+ cell count > 300/μL
Immunoglobulin (IgA) levels | Up to Day 360
Immunoglobulin (IgM) levels | Up to Day 360
T-cell Engraftment | Up to Day 360
  CD45 RA versus RO at 3, 6, 9 and 12 months
Disease-free survival | Two years
Incidence of secondary graft failure | Two years
Transplant-Related Mortality (TRM) | 100 Days
Quality of life using the World Health Organisation Five Wellbeing Index | Up to day 360
  QoL assessed at 3, 6, 9 and 12 months (World Health Organization [WHO] Five Wellbeing Index).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bacigalupo, MD, Principal Investigator — Unit for Hematology and BMT, Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy
Locations (2):
- University Hospital Centre Zagreb, Zagreb, Croatia
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No